CLINICAL TRIAL: NCT03040531
Title: Metabolic, Endocrine, and Central Effects of Genistein Aglycone in Glucocorticoid Induced Osteoporosis
Brief Title: Effects of Genistein Aglycone in Glucocorticoid Induced Osteoporosis
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Messina (Other)
Collaborators: Ministry of Health, Italy (Other Government)
Responsible Party: Principal Investigator, Francesco Squadrito, Full Professor of Pharmacology, University of Messina
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 45/16
Record Dates: First submitted 2017-01-30; First posted 2017-02-02 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2017-03

CONDITIONS: Osteoporosis, Steroid Induced
Keywords: glucocorticoid; genistein; alendronate
MeSH Terms: conditions — Osteoporosis | interventions — Alendronate; Calcium; Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Drugs will be labelled as "A" and "B" and so will be the groups. Patients and doctors involved will not be aware of the treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Genistein (Experimental): Each tablet will contain 27 mg of 98% pure genistein + 500mg Calcium + 200 IU Vit. D3. Subjects will receive 2 tablets per day 6 days/week for all the duration of the study.
  Once a week subjects will receive a tablet containing only 500mg Calcium + 200 IU Vit. D3.
  Interventions: Dietary Supplement: Genistein aglycone
- Alendronate (Active Comparator): Each tablet will contain 500mg Calcium + 200 IU Vit. D3. Subjects will receive 2 tablets per day 6 days/week for all the duration of the study.
  Once a week subjects will take one tablet containing 70mg alendronate.
  Interventions: Drug: Alendronate Oral Tablet; Dietary Supplement: Calcium + vitamin D3 tablet

INTERVENTIONS:
Dietary Supplement: Genistein aglycone — 27mg bid in tablets
  Other Names: fosteum
  Arms: Genistein
Drug: Alendronate Oral Tablet — 70 mg/week in tablets
  Other Names: Fosamax
  Arms: Alendronate
Dietary Supplement: Calcium + vitamin D3 tablet — 500mg Calcium + 200 IU Vitamin D3 bid in tablets
  Arms: Alendronate

SUMMARY:
Prolonged glucocorticoid therapy affects bone fragility, cardiovascular health, glucidic and lipidic metabolism, thyroid and brain function. Glucocorticoid-induced osteoporosis is characterized by low bone turnover and fractures, which occur in 30-50% of patients. Glucocorticoids affect predominantly cancellous or trabecular bone, increasing the risk of vertebral fractures, which may be asymptomatic and occur early during the first months of glucocorticoid treatment. Genistein exerts biological effects by several potential mechanisms. Besides protective effects on bone loss, genistein reduces cardiovascular risk markers, improves endothelial function and ameliorates glucose and lipid metabolism. This study is aimed at demonstrating genistein efficacy in glucocorticoid-induced osteoporosis in a cohort of caucasian post-menopausal women.

DETAILED DESCRIPTION:
Glucocorticoid-induced osteoporosis (GIOP) is one of the primary side effects of glucocorticoid use resulting in increased risk of fractures. Glucocorticoid therapy affects bone mass, glucidic and lipidic metabolism, thyroid function and is also responsible for a decline in cognitive function. In this study a natural approach will be used, a soy-derived isoflavone, namely genistein. Genistein has been proven effective in preserving bone mineral density in post-menopausal women, and has an high safety profile. Genistein was also able in improving cardiovascular markers, as well as lipidic and glucidic metabolism markers without interfering with thyroid function.

Treatment guidelines for the use of glucocorticoids have been established which advise that if prednisolone is administered at 5 mg per day for three months or longer requires regular monitoring of bone mineral density (BMD) and treatment to prevent osteoporosis must be initiated (American college of Rheumatology). Vitamin D and calcium are also recommended for the management of all patients treated with glucocorticoids. Bisphosphonates should be considered for the prevention and treatment of this disorder, because they can prevent the initial loss of bone mass from glucocorticoids. Alendronate, risedronate, and zoledronic acid were shown to prevent and reverse the loss of BMD in glucocorticoid-induced osteoporosis with greater effects than those observed with vitamin D and calcium. In fact, bisphosphonates induce improvement of BMD that is 2-fold greater than that observed during vitamin D treatment alone (4.6% vs. 2.0%, respectively). Anabolic therapy is also used for the treatment of glucocorticoid-induced osteoporosis. Teriparatide causes a greater increase in BMD than alendronate and greater reduction in the risk of vertebral fractures. Even with these evidentiary clinical trials and guidelines, patient bone loss is, in general, poorly managed. In glucocorticoid-induced osteoporosis, fractures also occur at higher BMDs than in postmenopausal osteoporosis in untreated women. Consequently, guidelines for the treatment of postmenopausal osteoporosis are not applicable to glucocorticoid-induced osteoporosis, and patients should be treated at BMD T-scores of -1.0 to -1.5 standard deviations. In addition, vertebral fractures may be asymptomatic and often require radiological diagnosis before treatment.

During the initial phases of glucocorticoid exposure bone resorption is increased. Glucocorticoids inhibit the formation of mature osteoblasts, but also activate an activate apoptosis in these cell types. Osteoprotegrin (OPG) expression, a key factor involved in modulating maturation of osteoclasts, is reduced also by glucocorticoids resulting in increased osteoclastogenesis. Therefore, the combination of reduced osteoblast formation, increased osteoclast maturation leads to accelerated bone loss while on glucocorticoid therapy. Therapies are needed which modulate osteoclast as well as osteoblast activity to restore a more normal balance to the bone remodeling process in glucocorticoid treated patients.

A rational treatment for glucocorticoid-induced osteoporosis should combine a significant anti-osteoporotic and anti-fracture activity with positive actions on the several undesirable effects of this therapy including alteration in glucose and lipid metabolism, amplification of the cardiovascular risk, impairment in thyroid and cognitive function.

Genistein aglycone represents an innovative therapeutic bullet to challenge the metabolic derangements induced by glucocorticoids. Among the anabolic compounds tested in recent years genistein aglycone seems a promising agent able to stimulate bone formation and to reduce bone resorption, acting via a genomic as well as a non-genomic pathways. Genistein is an isoflavone found in small quantities in certain legumes throughout the plant kingdom. Genistein has both ER agonist and antagonist activity in different cell types and works in a promoter specific manner in gene activation via ERs. Effects of genistein on bone metabolism derived from direct and indirect actions on bone cells and can be summarized in stimulation of osteoblastic bone formation and inhibition of osteoclastic bone resorption.

It has been demonstrated that genistein inhibits glucocorticoid receptor transactivation and may also induce a proteosomal degradation of the glucocorticoid receptor complex via the p53 and ubiquitin pathways. Another mechanism might involve genistein activity as a tyrosine kinase inhibitor via the limitation of the subcellular nuclear transport and the recycling of the glucocorticoid receptors, inhibiting in turn the effects of glucocorticoids on bone. In a rat model, we studied genistein preservative effects on methylprednisolone-induced bone loss and osteonecrosis of the femoral head. In our study genistein succeeded in preventing osteoporosis and osteonecrosis of the femoral head when co-administered with the glucocorticoid. The isoflavone statistically maintained bone mineral density and content over the methylprednisolone-treated group and showed comparable efficacy with the vehicle group. Genistein co-administered with methylprednisolone also statistically maintained femoral bone's resistance to rupture compared with the methylprednisolone group and preserved the normal architecture of cartilage as well as both cortical and trabecular bones with a well-organized matrix in femoral head.

Besides the protective effects on osteoporosis, genistein has been shown to positively affects the cardiovascular system reducing predictors of cardiovascular risk, improving endothelial function and ameliorating glucose and lipid metabolism. In addition genistein possesses beneficial activity in the central nervous system and protects the hippocampus from injury.

Regarding the effects of genistein on thyroid function that may be impaired by glucocorticoids a recent clinical trial evaluated the effects of three year administration of pure genistein aglycone (54 mg/day) on thyroid-related markers, in postmenopausal women. Specifically, changes in thyroid hormone receptors and thyroid hormone enzymes, blood levels of thyroid hormones and thyroid auto-antibodies were assessed. The results of this research showed that daily consumption of genistein aglycone did not modified circulating fT4 (free thyroxine), fT3 (free triiodothyronine), and TSH (thyroid-stimulating hormone) levels; further, genistein aglycone administration over 3 yr did not affect the enzymes involved in thyroid hormone production, the thyroid hormone auto-antibodies, and the expression of thyroid hormone receptors then confirming that genistein does not appear to alter thyroid function in postmenopausal women.

Taken together this clinical and pre-clinical observations lead the investigators to hypothesize a role for genistein in the management of glucocorticoid-related side effects.

ELIGIBILITY:
Inclusion Criteria:

* being treated with glucocorticoids (5 mg of prednisone equivalents) for the preceding 3 months or less, and expect to continue the therapy for at least 12 months;
* being post-menopausal;

Exclusion Criteria:

* use of other steroids or osteoporosis medications;
* have been diagnosed with metabolic bone diseases (other than glucocorticoid osteoporosis)
* previous (1 year) or current use of HRT (hormone replacement therapy)
* other diseases that may affect participation (i.e. mental illness)

Ages: 54 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Only female XX patients will be included, to avoid interactions with other steroid drugs.
Enrollment: 200 (Estimated)
Dates: Start 2017-01-19 (Actual); Primary Completion 2018-06-30 (Estimated); Study Completion 2018-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in Bone mineral density | 24 months
  BMD of lumbar spine and femoral will be measured by DEXA (dual energy x-ray absorptiometry)
Bone fracture | 24 months
  Xrays of the lumbar spine (T4-L4) will be taken to evaluate the presence of fractures
Change in Bone quality | 24 months
  pQCT (peripheral quantitative computed tomography) will be used for bone quality evaluation

SECONDARY OUTCOMES:
Change in Bone markers | 24 months
  bone turnover markers will be evaluated on peripheral blood
Change in Cardiovascular markers | 24 months
  Markers of cardiovascular risk will be evaluated on peripheral blood
Change in Glucose and lipid metabolism | 24 months
  Glycaemia and blood lipids will be evaluated on peripheral blood
Change in Quality of life | 24 months
  European Quality of Life Questionnaire will be administered to subjects
Chage in skin elasticity | 24 months
  skin elasticity will be tested in subjects taking glucocorticoids
Change in thyroid markers | 24 months
  markers of thyroid function will be evaluated on peripheral blood
Change in inflammatory markers | 24 months
  markers of inflammation will be evaluated on peripheral blood
Polymorphisms of estrogen receptor | 24 months
  Estrogen receptor polymorphisms will be evaluated on white blood cells

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Squadrito, MD, Study Director — University of Messina
Locations (2):
- Italy (2):
  - University of Messina, Messina, Italy
  - University Hospital, Messina

IPD SHARING:
Plan to Share IPD: No